CLINICAL TRIAL: NCT04276259
Title: Neurocomputational Mechanisms of Mood Improvement
Brief Title: Rapid Antidepressant Improvement Secondary to Excitatory Brain Responses
Acronym: RAISE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marta Peciña, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Marta Peciña, MD PhD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: STUDY19050307
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Buprenorphine; Naltrexone

STUDY DESIGN:
Intervention Model Description: This is a mechanistic trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Buprenorphine Injection + Oral Placebo Pill (Experimental): Buprenorphine is a μ-opioid partial agonist and kappa-opioid antagonist that is used to treat moderate to severe pain and opioid dependence. The intramuscular administered opioid agonist which will be used to modulate reward learning signals to understand placebo effects in patients with depression. In the buprenorphine condition, participants will receive one IM injection of 0.3mg/1ML buprenorphine hydrochloride (Buprenex®. Richmond, VA: Reckitt Benckiser Pharmaceuticals Inc.; 2006) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~6 hours) and an oral placebo tablet.
  Interventions: Drug: Buprenorphine; Drug: Oral Placebo; Device: Theta burst stimulation (TBS) of the ventromedial prefrontal cortex.
- Naltrexone Oral Tablet + Intramuscular Saline Injection (Experimental): Naltrexone is thought to strongly block μ-opioid receptors. Oral (pill) opioid antagonist which will be used to modulate reward learning signals to understand placebo effects in participants with depression. In the naltrexone condition, participants will receive one tablet of 50mg Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours) and a saline IM injection.
  Interventions: Drug: Naltrexone; Drug: IM Placebo; Device: Theta burst stimulation (TBS) of the ventromedial prefrontal cortex.
- Oral Placebo Pill + Intramuscular Saline Injection (Experimental): Inert pill and saline injection that have no inherent power to produce an effect. In the inert pill condition, participants will receive one IM arm injection of saline (1ML) and an oral placebo tablet.
  Interventions: Drug: Oral Placebo; Drug: IM Placebo; Device: Theta burst stimulation (TBS) of the ventromedial prefrontal cortex.

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine is a μ-opioid partial agonist and kappa-opioid antagonist that is used to treat moderate to severe pain and opioid dependence. The intramuscular administered opioid agonist which will be used to modulate reward learning signals to understand placebo effects in patients with depression. In the buprenorphine condition, participants will receive one IM injection of 0.3mg/1ML buprenorphine hydrochloride (Buprenex®. Richmond, VA: Reckitt Benckiser Pharmaceuticals Inc.; 2006) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~6 hours) and an oral placebo tablet.
  Arms: Buprenorphine Injection + Oral Placebo Pill
Drug: Naltrexone — Naltrexone is thought to strongly block μ-opioid receptors. Oral (pill) opioid antagonist which will be used to modulate reward learning signals to understand placebo effects in participants with depression. In the naltrexone condition, participants will receive one tablet of 50mg Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours) and a saline IM injection.
  Arms: Naltrexone Oral Tablet + Intramuscular Saline Injection
Drug: Oral Placebo — Oral placebo: to match the oral naltrexone.
  Arms: Buprenorphine Injection + Oral Placebo Pill; Oral Placebo Pill + Intramuscular Saline Injection
Drug: IM Placebo — IM saline placebo: to match the i.v. buprenorphine.
  Arms: Naltrexone Oral Tablet + Intramuscular Saline Injection; Oral Placebo Pill + Intramuscular Saline Injection
Device: Theta burst stimulation (TBS) of the ventromedial prefrontal cortex. — Participants will receive two blocks of each TBS form. During the first block, stimulation intensity will be gradually escalated in 5% increments (from 80% to 110% rMT) in order to enhance tolerability. In all conditions, the investigators will apply 600 pulses of theta burst at 110% RMT. Each block of iTBS will consist of 20 trains, each lasting 2s with intertrain intervals of 8s, for a total of 192s. Each block of cTBS will consist of one continuous train of 40s. The sTBS will make use of two surface electrodes placed on the scalp.
  Other Names: sham (s), continuous (c) and intermittent (i).

SUMMARY:
The central goal of this application is to demonstrate the causal contribution of reward learning signals (expected values and reward prediction errors [RPE]) to antidepressant responses (Aim1) by experimentally manipulating expected values using transcranial magnetic stimulation (TMS) targeting the vmPFC (Aim 2) and μ-opioid striatal RPE signal using pharmacological approaches (Aim 3).

DETAILED DESCRIPTION:
The central goal of this study is to demonstrate the causal contribution of reward learning signals (expected values and RPEs) to antidepressant responses (Aim1) by experimentally manipulating expected values using transcranial magnetic stimulation (TMS) targeting the vmPFC (Aim 2) and μ-opioid striatal RPE signal using pharmacological approaches (Aim 3). In a 3x3 factorial double-blind trial, the investigators will randomize 120 unmedicated major depressive disorder (MDD) adults (18-55 years) to one of three between-subject opioid conditions: the μ-opioid agonist buprenorphine (n=40), the μ-opioid antagonist naltrexone (n=40), or the inert pill (n=40). Within each arm, individuals will be assigned to receive three within-subject counterbalanced sessions of TMS targeting the vmPFC-intermittent TBS (iTBS) expected to potentiate the vmPFC, continuous TBS (cTBS) expected to de-potentiate the vmPFC, and sham TBS (sTBS). These experimental manipulations will be used to modulate trial-by-trial reward learning signals and related brain activity during the Antidepressant fMRI Task. Understanding the mechanisms underlying antidepressant responses is essential to identify novel therapeutic targets for depression.

ELIGIBILITY:
Inclusion Criteria:

* • Adults, age 18-55 years; fluent in English and with the capacity to understand the nature of the study and sign the written informed consent since the research instruments used in this study are not available in other languages;

  * Written informed consent obtained;
  * A score on the Mood and Anxiety Symptom Questionnaire- Anhedonic Depression (MASQ-AD) ≥ 23 (2/3 sample) and MASQ-AD < 23 (1/3 sample) with or without certain anxiety disorders (e.g., generalized anxiety, panic, agoraphobia, social phobia, and specific phobia);
  * No more than one failed antidepressant trial of adequate dose and duration, as defined by the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ);
  * Participants can have previous history of antidepressant treatment but will need to be antidepressant medication-free for at least 21 days prior to the collection of imaging data (five weeks for fluoxetine).

Exclusion Criteria:

* • Pregnant or breastfeeding or plan to become pregnant over the duration of the study;

  * History (lifetime) of psychotic depressive, schizophrenic, bipolar (I, II, or NOS), schizoaffective, or other Axis I psychotic disorders;
  * Meeting M.I.N.I. criteria for substance dependence in the last 6 months, except for nicotine, or substance abuse in the last 2 months;
  * Requiring immediate hospitalization for psychiatric disorder or have an unstable general medical condition (GMC) that will likely require hospitalization or to be deemed terminal (life expectancy < 6 months after study entry);
  * Having epilepsy or other conditions requiring an anticonvulsant;
  * Receiving vagus nerve stimulation, electroconvulsive therapy, or repetitive Transcranial Magnetic Stimulation during the current episode.
  * Currently taking any psychiatric medication or other potential augmenting agents (e.g., T3 in the absence of thyroid disease, lithium, buspirone); Taking thyroid medication for hypothyroidism may be included only if they have been stable on the thyroid medication for 3 months;
  * Receiving therapy that is depression specific, such as Cognitive Behavioral Therapy or Interpersonal Psychotherapy of Depression (participants can participate if they are receiving psychotherapy that is not targeting the symptoms of depression, such as supportive therapy, marital therapy);
  * Currently actively suicidal or considered a high suicide risk;
  * Patients are receiving opioid analgesics.
  * Patients are currently dependent on opioids.
  * Patients are in acute opioid withdrawal.
  * Any individual who has failed the naloxone challenge test or who has a positive urine screen for opioids.
  * Any individual with a history of sensitivity to buprenorphine or naltrexone.
  * Currently enrolled in another study, and participation in that study contraindicates participation in this study;
  * Any reason not listed herein yet, determined by the site PI and research staff that makes participation in the study hazardous.
  * Having any contraindication for the performance of TMS, such as the presence of a neurologic disorder or medication therapy known to alter seizure threshold (e.g., stroke, aneurysm, brain surgery, structural brain lesion, brain injury, frequent/severe headaches), recurrent seizures or epilepsy in participant or family history of hereditary epilepsy, pregnancy, metallic implants in body or other devices that may be affected by magnetic field or significant heart disease or cerebrovascular disease.
  * Having any contraindication for the performance of an MRI, such as the presence of metal implants or foreign metallic objects (e.g., braces or extensive dental work), severe claustrophobia, or inability to tolerate the scanning procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
BOLD Responses in the vmPFC-VS circuit | Approximately at day 7, 14, 21.
  Changes in blood oxygenation level-dependent (BOLD) signal during the Antidepressant fMRI Task.
TBS Effects of BOLD Response | Approximately at day 7, 14, 21.
  Changes in BOLD signal during the Antidepressant fMRI Task between iTBS vs. sTBS, and cTBS vs. sTBS.
Opioid Modulation Effects on BOLD Responses in the vmPFC-VS circuit | Approximately at day 7, 14, 21.
  Changes in BOLD signal during the Antidepressant fMRI Task between Buprenorphine vs. inert pill, and Naltrexone vs. inert pill.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Peciña, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bellefield Tower, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with NIMH Data Archive (NDA) policies, the investigators will obtain relevant GUIDs and experiment IDs in order to upload all relevant data biannually. The investigators will use the Validation and Upload Tool for CSV files from behavior during the fMRI experiment, and NIfTI-formatted images for imaging. The investigators will upload study data cumulatively every 6 months per NDA guidelines, with the exception of imaging data, which are will be uploaded in installments.
  The final research data will not contain any identifiable information and will be deposited in the Research Domain Criteria Database (RDoCdb) repository in the NDA prior to the acceptance for publication of the main findings from the final dataset. Documentation and code for computational models developed as part of this project will be shared via a Github page (https://github.com/).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Pecina M, Dombrovski AY, Price R, Karim HT. Understanding the Neurocomputational Mechanisms of Antidepressant Placebo Effects. J Psychiatr Brain Sci. 2021;6:e210001. doi: 10.20900/jpbs.20210001. Epub 2021 Feb 15. PMID 33732892